CLINICAL TRIAL: NCT06450756
Title: Effect of Male Involvement in Family Planning Education on Contraceptive Use Among Married Couples in the Pastoralist Community of Fentale District, Eastern Ethiopia.
Brief Title: Effect of Male Involvement in Family Planning Education on Contraceptive Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jimma University (Other)
Responsible Party: Principal Investigator, Sena Adugna Beyene, Senior Lecturer of Statistics, Population studies(Reproductive Health), and Public Health Senior Researcher, Jimma University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: SAB2019
Record Dates: First submitted 2024-06-05; First posted 2024-06-10 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Contraceptive Usage; Family Planning
MeSH Terms: conditions — Contraception Behavior

STUDY DESIGN:
Who Masked: Participant
Masking Description: Only the study participants were masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Couples arm . (Experimental): The Couples Arm intervention addressed gaps identified from baseline findings. It involved comprehensive family planning education delivered to married women and men by community agents, Health Extension Workers, and FP experts using flyers, booklets, and face-to-face discussions. Health Extension Workers supported community agents in delivering health education messages about family planning twice a month for 6 months, with each session lasting 2 hours. Note: The group size for the Couples Arm was 748 couples (374 women and 374 men).
  Interventions: Behavioral: Couples arm
- Male arm (Experimental): The intervention in the married male arm provided health education based on baseline findings to address gaps. Community agents and videos featuring men involved in family planning (FP), a male model supporting his wife's FP use, and a supportive husband sharing information with his wife were used. Clan leaders "Abbaa Gada" (Indigenous Oromo), religious leaders, and district FP experts also played key roles. Monthly 1-hour sessions over 6 months delivered health education messages about FP. The 374 men selected were the husbands in the intervention group, participating in household and individual-level interventions alongside their wives and attending community gatherings twice. Note: The group size for the male arm (Male Involvement group) was 374 men.
  Interventions: Behavioral: Male arm
- Control arm (No Intervention): This arm of the Couples-based intervention involves observing the community without providing male education or couples' education at the household/individual level. There is no active intervention by the researchers, but government family planning activities continue. Couples in the control arm are not exposed to the comprehensive interventions of the intervention arms. They only receive the standard intervention as per national guidelines, involving routine reproductive health care. 748 couples (374 women and 374 men) were assigned to the control group, with routine healthcare access or no specific intervention. Note: The group size for the control arm was 748 couples (374 women and 374 men).

INTERVENTIONS:
Behavioral: Couples arm — The Couples Arm aims to improve family planning (FP) utilization in pastoralist communities, addressing significant disparities in contraceptive use and unmet FP needs between pastoralist and agrarian communities in Ethiopia. Pastoralist areas face challenges such as low contraceptive usage, high unmet FP needs, and elevated rates of maternal and child morbidity and mortality. In 2016, only 9.1% of women in pastoralist areas used contraceptives, compared to a 41% prevalence rate in 2019 for the general population in Ethiopia. Reasons for non-use of contraceptives include lack of knowledge, unwillingness, negative perceptions, desire for many children due to child mortality concerns, and male dominance in FP decision-making. The study hypothesizes that engaging men and educating women about FP could enhance FP utilization, increase male involvement in family planning, and empower women.
  Other Names: Women Empowerment.
  Arms: Couples arm .
Behavioral: Male arm — This arm focused on promoting male involvement in family planning (FP) through comprehensive health education and video messages. Husbands were encouraged to become supportive partners and share FP information with their wives. Separate education sessions were held for men, recognizing their greater exposure to social activities and information in pastoralist contexts. Pastoralist wives typically rely on their husbands for information due to limited social access. Women in pastoral communities have significant informal power in family decisions, influenced by factors such as age, husband's status, sons' ages, eloquence, and wisdom. Reproductive health discussions are primarily between husband and wife. Education aimed to improve modern contraceptive use, overcoming common barriers like husband objection and religious influence on decision-making.
  Other Names: Male Involvement Arm
  Arms: Male arm

SUMMARY:
This study aimed to examine the effect of Male Involvement in Family Planning Education on Contraceptive Use Among Married Couples in the Pastoralist Community of Fentale District, Eastern Ethiopia.

DETAILED DESCRIPTION:
The rationale for conducting this study stemmed from the persistent challenges in family planning (FP) utilization observed within pastoralist communities, particularly in the Fentale District of Eastern Ethiopia. Despite progress in modern contraceptive use and male involvement in FP at the national level, these communities continue to face limited male involvement in Family planning and contraceptive coverage. Therefore, the study aimed to address this issue by implementing an integrated behavioral model through a quasi-experimental design. The objective was to assess the effectiveness of various intervention approaches, including strategies to increase male involvement and household-based education, in improving FP utilization among couples in the Fentale District. This evaluation was deemed crucial to address the ongoing challenges and increase contraceptive uptake in pastoralist regions. Fentale District was selected exclusively for this study due to several criteria, including accessibility, social structure, economic strength, and its pastoralist nature. These factors made it an ideal location to examine the impact of interventions on FP utilization within pastoralist communities. In a quasi-experimental study conducted in Fentale District, Eastern Ethiopia, 1496 married couples (748 controls, 748 interventions) were selected through systematic random sampling. Among them, 748 couples (comprising 374 women and 374 men) were assigned to the intervention group. Simultaneously, the remaining 748 couples (also comprising 374 women and 374 men) were assigned to the control group and received routine healthcare access or no specific intervention. It's noteworthy that the 374 men selected for the study were the same individuals as the husbands in the intervention group, participating in household-level or individual-level interventions alongside their wives. Additionally, these men were also part of the Male Involvement Arm, attending community gatherings for a second time, thereby ensuring their participation in both arms of the study.

ELIGIBILITY:
Inclusion Criteria:

* Married women aged between 15 and 49 years, along with their husbands.
* Non-pregnant women at the time of the study period were included, along with their husbands.
* Only legally married couples were considered.
* Couples who have resided in the village or an area with consistent mobility for the past year.
* Couples cohabiting in the same house within the study area or in areas with mobility were included.
* Couples intending to stay in the district or areas with mobility for at least one year and six months from the data collection period.
* Inclusion of couples where the husband expressed willingness for his wife to participate in the study.
* Only mentally capable couples, ensuring individuals without cognitive impairments, were part of the research.
* Husbands within monogamous marriages (having only one wife) were eligible for analysis.
* Written informed consent was obtained from husbands on behalf of wives under 18, respecting the cultural context and norms of the study area.

Exclusion Criteria:

* Married women not within the reproductive age range (15-49 years old) were excluded from the study, along with their husbands.
* Not Legally married Couples excluded.
* Couples where the husband was unwilling to include his wife in the study were excluded. - Mentally incapable couples, indicating those with cognitive impairments, were not considered in the study.
* Husbands within polygamous marriages (having more than one wife) were also excluded from the analysis, aiming to streamline the focus on monogamous marital dynamics.
* Pregnant women at the time of the survey, along with their husbands were excluded.
* Couples who had not resided in the village or areas with mobility. For the past year were excluded.
* Couples not cohabiting in the same house in the study area or areas with mobility. Were excluded.
* Those who did not plan to stay in the district area or areas with mobility for at least one year and six months from the time of data collection were excluded.
* These exclusions were implemented to enhance the clarity of the study's focus and minimize redundancy of information

Ages: 15 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Participants self-identifying as male were included in the evaluation to assess male involvement in family planning decision-making and support.
Enrollment: 1496 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-06-27 (Actual); Study Completion 2022-07-03 (Actual)

PRIMARY OUTCOMES:
Contraceptive Utilization Rate | Up to six months
  The contraceptive utilization rate was assessed among the study participants. The proportion of married couples who used the contraceptive was compared using the baseline and end-line data from the intervention.

SECONDARY OUTCOMES:
Men Involvement in Family planning | Up to six months
  The evaluation of male involvement over the 6-month intervention from January 1 to July 3, 2022, was part of the secondary outcome measures. This assessment, conducted at 6 months, utilized a set of 10 items: 3 focused on couples' discussions about family planning (FP) and 7 on husbands' support for their wives. Topics included discussing FP, birth spacing, and limiting births. Spousal support actions assessed included accompanying to health facilities, participating in FP choices, allowing FP use, reminding of schedules, assisting in domestic activities, providing financial support, and being aware of FP side effects. Perspectives on current and future FP support were gathered from both husbands and wives, including both current and non-users of contraception. This allowed for a comprehensive understanding of male involvement in FP decision-making.

CONTACTS AND LOCATIONS:
Overall Officials: Tefera Belachew, PhD, Study Chair — Jimma University; *, Sileshi Garoma, PhD, Study Chair — Departments of Public Health, Adama Hospital Medical College, Adama, Ethiopia
Locations (1):
- Jimma University, Jimma, Oromiya, Ethiopia

IPD SHARING:
Plan to Share IPD: No